CLINICAL TRIAL: NCT00002021
Title: An Open Study of Foscarnet Treatment of Acyclovir-Resistant Herpes Simplex Virus in Patients With the Acquired Immunodeficiency Syndrome and Other Immunodeficiencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astra USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 020F; 89-FOS-09A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-10

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Immune Tolerance; Injections, Intravenous; Herpes Simplex; Immunity, Cellular; Foscarnet; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — Herpes Simplex; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
To evaluate the safety and efficacy of intermittent intravenous (IV) foscarnet in the treatment of acyclovir-resistant herpes simplex virus (HSV) infections in AIDS patients and other immunocompromised patients. To evaluate the necessity, efficacy, and safety of IV maintenance foscarnet therapy in preventing recurrent disease. To confirm the pharmacokinetics of intermittent induction and maintenance IV regimens.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Cyclosporine.

Patients must have AIDS as defined by the CDC or be immunocompromised (transplant patients; other hematologic malignancies with recognized cell-mediated immune deficiency). Patients must also have herpes simplex virus (HSV) infection documented by culture and in vitro resistance to acyclovir by standard laboratory susceptibility or suspected resistance to acyclovir after an acyclovir treatment failure in which acyclovir was administered for at least 2 weeks intravenously at doses of 30 mg/kg/day (or a comparative dose adjusted for renal insufficiency). In vitro susceptibility data must be pending in the latter case. Patients must be able to give informed consent. Patients < 18 years of age may participate with the consent of parent, guardian, or person with power of attorney, or through the provisions of state laws regarding emancipated minors. Patients must have expected survival of at least 6 months.

Prior Medication:

Allowed:

* Cyclosporin.
* Ganciclovir.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Known allergy to foscarnet.
* Any clinically significant pulmonary or neurologic impairment (e.g., patients who are intubated or comatose).

Concurrent Medication:

Excluded:

* Any potentially nephrotoxic agent (except cyclosporine).
* Immunomodulators.
* Biologic response modifiers.
* Investigational agents.

Patients with the following are excluded:

* Known allergy to foscarnet.
* Any clinically significant pulmonary or neurologic impairment (e.g., patients who are intubated or comatose).

Prior Medication:

Excluded within 7 days of study entry:

* Any potentially nephrotoxic agent (except cyclosporin).
* Immunomodulators.
* Biologic response modifiers.
* Investigational agents.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA CARE Ctr, Los Angeles, California
  - Huntington Memorial Hosp, Pasadena, California

REFERENCES:
- [Background] Balfour HH Jr, Benson C, Braun J, Cassens B, Erice A, Friedman-Kien A, Klein T, Polsky B, Safrin S. Management of acyclovir-resistant herpes simplex and varicella-zoster virus infections. J Acquir Immune Defic Syndr (1988). 1994 Mar;7(3):254-60. PMID 8106965